CLINICAL TRIAL: NCT07315464
Title: Effects of Mobilization With Movement Versus Sustained Mobilization Along With Eccentric Exercises on Pain & Functional Disability in Patients With Knee Osteoarthritis
Brief Title: Effects of MWM Vs Sustained Mobilization on Knee Osteoarthritis
Acronym: MWM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCPT/DPT/ERB/35 FAKIHA
Record Dates: First submitted 2025-12-08; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Mobilization with Movement (MWM); Sustained Mobilization; Eccentric Exercises; Kellgren-Lawrence (KL) system; Numeric Pain Rating Scale (NPRS); Knee Injury and Osteoarthritis Outcome Score (KOOS)
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Intervention Model Description: This study follows a Randomized Controlled Trial (RCT) model designed to compare the effectiveness of Mobilization with Movement (MWM) and Sustained Mobilization (Kaltenborn), each combined with eccentric exercises, in patients with Grade III knee osteoarthritis. Participants will be randomly allocated into two intervention groups using a computer-generated sequence with block randomization to ensure equal group sizes. A single-blinded approach will be used, where participants will unaware of group assignment, while outcome assessments were performed by an independent blinded evaluator. This model allows controlled comparison of both mobilization techniques on pain reduction, functional improvement, and range of motion.
Who Masked: Outcomes Assessor
Masking Description: This study used a single-blinded design. Participants will be blinded to group allocation to minimize performance bias. Group assignment will be concealed through sealed, opaque, sequentially numbered envelopes, opened only after baseline assessment by an independent physiotherapist. The treating therapist will not be blinded due to the nature of manual therapy interventions. However, all outcome measurements-including pain, disability, and range of motion will be recorded by a separate blinded assessor to reduce detection bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan Mobilization (Experimental): This group will hold intervention for MWM including passive glides while the eccentric exercises includes slow controlled squats
  Interventions: Other: mulligan moblization
- Kaltenborn Mobilization (Active Comparator): This arm's intervention includes grade II traction and eccentric loading
  Interventions: Other: kaltenborn moblization

INTERVENTIONS:
Other: mulligan moblization — This group will receive total 3 sessions / week (9-12 sessions) Intensity includes Accessory Glide with pain free active knee motion + moderate intensity eccentric loading Type includes Mulligan MWM ( Passive Glide during active knee flexion/extension + Eccentric Quadricpes Exercises (Slow Controlled Squats ) Time 30-45 mins
  Other Names: slow controlled squats
  Arms: Mulligan Mobilization
Other: kaltenborn moblization — This group will receive frequency of 3 session/ week (9-12 sessions) Intensity includes Kaltenborn Grade II Traction according to pain tolerance + Moderate Intensity Eccentric Loading Type of Exercise includes Sustained Joint Mobilization in loose pack position + Quadriceps Exercises (Slow step down ) Time 35-45 mins
  Other Names: Eccentric Loading
  Arms: Kaltenborn Mobilization

SUMMARY:
This article focused on people diagnosed with grade III Knee OA with sample size of 68 patients , who will randomly divided into two groups . Group A received Mulligan's MWM while group B received Kaltenborn's Sustained Mobilization along with eccentric exercises. The goal of the study was to compare the effectiveness of these two treatment conditions in reducing knee pain and improving joint function decreasing disability in daily activities. The patients followed a structured treatment plan over a set period and outcomes will measured using reliable clinical tools such as NPRS for pain KOOS for functional disability and Goniometer for ROM.

DETAILED DESCRIPTION:
The word osteoarthritis (OA) is comprised of two separate terms: the prefix "osteo" means bone, and arthritis means joint inflammation. Subcommittee on Osteoarthritis of the American Rheumatism Association, Diagnostic and Therapeutic Criteria Committee, defined OA as "a heterogeneous group of conditions that lead to joint symptoms and signs which are associated with defective integrity of articular cartilage, in addition to related changes in the underlying bone and at the joint margins. "The prevalence of knee pain and symptomatic OA is double in female as compared to male over 20 years. According to a study in people of age 45 or above prevalence of OA is 20% in women and 10% in men. The causes of knee OA include factors such as age, gender, weight, genetics, injuries, and overuse. Common signs and symptoms of knee OA include knee pain, joint stiffness, decreased muscle strength, and proprioceptive deficits. In addition, individuals with knee OA often exhibit poor neuromuscular control, slower walking speed, decreased functional ability, and an increased susceptibility to falling.The most common scale for knee OA classification is the Kellgren-Lawrence (KL) system, which evaluates osteophyte formation, articular cartilage narrowing associated with subchondral bone sclerosis, and altered shape of bone ends from grade 0 to grade 4.

KL classification:

Grade 0: no narrowing; Grade 1: doubtful articular space constriction, osteophytic lipping is possible; Grade 2: permanent osteophytes, potential constriction of the joint space; Grade 3: mild osteophytes, definite constriction of the joint space, and potential end-bone deformation; Grade 4: severe osteophytes, severe constriction of the joint space, severe sclerosis, and definite deformation of the bone.

Radiographes or X-rays to assess pain and restlessness are the foundation for detecting and diagnosing knee OA. Key features that can be observed using X-rays are joint space narrowing, osteophytes, cyst formation, and subchondral sclerosis.The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a wellknown useful diagnostic tool to assess knee ligament injury and osteoarthritis. It includes 42 items in five sub-scales evaluating pain, symptoms, function of daily living, sport and recreation function (sport/rec), and (QOL).The Management of knee OA needs a multidisciplinary approach. The conservative treatment forms for knee OA comprise pharmacological and non-pharmacological modalities. Non-steroidal anti-inflammatory drugs (NSAIDS) are mostly used for pain relief and stiffness caused by OA, with the numerous side effects, particularly on the gastrointestinal tract, making the treatment unsustainable.Manual therapy is a technique used to treat musculoskeletal dysfunctions and pain and usually includes manual therapies, such as massages, joint mobilization, and manipulations. Among the mobilization techniques, Mulligan's mobilization with movement (MWM) has been considered a good alternative for the treatment of musculoskeletal disorders, improving pain and ROM.MWM is based on the concept that minor position faults occur in articulating surfaces of joints following injury or strains, resulting in movement restriction and pain exacerbated by active contraction of muscles within the faulty positions of the joint. Thus, MWM involves passive accessory glide as a corrective technique, applied by the therapist perpendicular to the joint plane to correct the positional fault, combined with the offending movement being performed actively by the subject and sustained for several repetitions. The pain should always be reduced and/or eliminated during the application, and pain-free function should be restored.Sustained mobilisation is a hands-on therapy technique often used in the treatment of knee OA to help reduce pain and improve how well the joint moves. It involves gently holding the joint in a stretched or distracted position for a period of time, which can help loosen stiff tissues, improve joint lubrication, and ease discomfort. For people with knee osteoarthritis-who often experience pain, stiffness, and limited mobility-this type of mobilisation can be a useful way to manage symptoms and support better function. When combined with exercises and other rehabilitation strategies, sustained mobilisation may play a valuable role in improving overall joint health and quality of life.Eccentric exercise actions are characterized by low energy cost, high force production, hypertrophic impact, and a favorable effect on fall risk, physical function, and mobility. Eccentric resistance training may also increase volitional drive and reduce corticospinal inhibition to the muscle more than concentric training in OA. Eccentric actions are essential in daily activities, such as stair descent, squatting, or sitting into a chair.Therefore, this study aims to directly compare MWM and sustained mobilization, each integrated with eccentric strengthening exercises, to determine which approach is more effective for improving pain, range of motion, and functional performance in patients with Grade 3 knee OA. The findings will support physiotherapists in selecting the most appropriate, evidence-based interventions to enhance quality of life and functional independence for individuals living with moderate knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

Age between 45 and 70 years Both male and female patients with a history of knee osteoarthritis were selectedfor this study. Clinically and radiologically diagnosed with Grade III Knee Osteoarthritis (basedon Kellgren and Lawrence scale).

Meets ACR criteria for knee OA

Exclusion Criteria:

History of knee or lower limb surgery Received corticosteroid injections (oral or intra-articular) in the past 6 months Other musculoskeletal conditions in the lower limb(e.g., fracture, bursitis, back pain with radiating symptoms) Diagnosed with inflammatory joint diseases (e.g., rheumatoid arthritis, gout) Neurological conditions affecting lower limbs (e.g., stroke, neuropathy) BMI > 35 (severe obesity) that limits safe participation in exercises Any contraindications to manual therapy (e.g., malignancy, infection, unstablejoint)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  The tool used for accessing pain is NPRS. The Numeric Pain Rating Scale (NPRS) is a widely used subjective measure for assessing pain intensity, where participants rate pain on a scale from 0 to 10. A score of 0 indicates no pain, while 10 represents the worst pain imaginable. The NPRS is simple, quick to administer, and highly useful for tracking changes in pain levels over time, evaluating treatment effectiveness, and guiding clinical decision-making. Its reliability and ease of use make it a standard tool in both clinical practice and research settings. Both MWM and Sustained Mobilization aim to reduce pain. The time frame for assessing pain is 4 weeks . While investigator aim to measure at baseline , week 2 and week 4 .
Functional Disability | 4 weeks
  The tool used for accessing functional disability is KOOS. The KOOS is a comprehensive, patient-reported outcome measure used to evaluate symptoms, functional limitations, and quality of life in individuals with knee injuries or knee osteoarthritis. It includes five subscales: Pain, Symptoms, Activities of Daily Living (ADL), Sport and Recreation Function, and Knee-related Quality of Life. Each item is scored on a 5-point Likert scale and then converted to a 0-100 scale, where 0 represents extreme knee problems and 100 indicates no knee problems. Each subscale is scored independently, allowing clinicians and researchers to assess specific domains of knee function and monitor changes over time. The KOOS is valued for its sensitivity to both short-term and long-term functional outcomes. While invesyigator aim to measure at baseline , week 2 and week 4 .

SECONDARY OUTCOMES:
ROM | 4 weeks
  The tool used for accessing ROM is Goniometer. A goniometer is a standard clinical tool used to measure the range of motion (ROM) in patients with knee osteoarthritis. It provides an objective assessment of joint mobility by measuring angles during knee flexion and extension. The stationary arm is aligned with the femur, the movable arm with the tibia, and the axis is positioned over the lateral epicondyle of the femur. ROM values help identify functional limitations, monitor disease progression, and evaluate the effectiveness of therapeutic interventions. Accurate goniometric measurement is essential for documenting baseline impairments and tracking improvements throughout rehabilitation.The time frame for assessing pain is 4 weeks . While investigator aim to measure at baseline , week 2 and week 4 .

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo hospital, Ghurki Trust Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent KR, Vincent HK. Concentric and Eccentric Resistance Training Comparison on Physical Function and Functional Pain Outcomes in Knee Osteoarthritis: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2020 Oct;99(10):932-940. doi: 10.1097/PHM.0000000000001450. PMID 32324615
- [Background] Heidari B. Knee osteoarthritis prevalence, risk factors, pathogenesis and features: Part I. Caspian J Intern Med. 2011 Spring;2(2):205-12. PMID 24024017
- [Background] Kataria Sweta Shah, K., Effect of Kaltenborn Traction versus Mulligan Mobilization with Movement as an adjunct to Conventional Exercise on Pain and Functions in Knee Osteoarthritis. International Journal of Science and Research (IJSR), 2023. 12(3): p. 1178-1182.
- [Background] Gul, H. and I. Tahir, EFFECTS OF MULLIGAN ROTATIONAL MOVEMENT VERSUS MEDIAL GAPPING TECHNIQUE ON PAIN, RANGE OF MOTION AND DISABILITY IN PATIENTS WITH KNEE OSTEOARTHRITIS. Pakistan Journal of Rehabilitation, 2024. 13(1): p. 99-110.